CLINICAL TRIAL: NCT02324738
Title: Open-Label Study to Evaluate Potential Pharmacokinetic and Pharmacodynamic Interactions of Orally Administered Mefloquine and Dihydroartemisinin-Piperaquine in Healthy Adult Subjects
Brief Title: Pharmacokinetic and Pharmacodynamic Study of Mefloquine and Dihydroartemisinin-Piperaquine in Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMEC 14-069
Record Dates: First submitted 2014-12-15; First posted 2014-12-24 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: Mefloquine/Dihydroartemisinin-piperaquine; drug interaction
MeSH Terms: interventions — Mefloquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy Volunteer (Experimental): All subjects will receive Mefloquine and Dihydroartemisinin-piperaquine, wash out then will receive Mefloquine
  Interventions: Drug: Mefloquine and Dihydroartemisinin-piperaquine; Other: Wash-out period; Drug: Mefloquine

INTERVENTIONS:
Drug: Mefloquine and Dihydroartemisinin-piperaquine — 2 tablets of mefloquine and 3 tablets of dihydroartemisinin-piperaquine single dose
Other: Wash-out period
Drug: Mefloquine — 2 tablets of Mefloquine single dose

SUMMARY:
This is an open-label sequential pharmacokinetic study in 16 healthy glucose-6-phosphate dehydrogenase (G6PD) normal Thai subjects at Faculty of Tropical medicine, Mahidol university.

The 16 subjects have already participated in a healthy volunteer studies in the past either i) Open-Label Study to Evaluate Potential Pharmacokinetic Interaction of Orally Administered primaquine and dihydroartemisinin-piperaquine (DHA-PQP) in Healthy Adult Subjects or ii) Comparison of the electrocardiographic effects in relation to Pharmacokinetic profile of chloroquine and piperaquine in healthy Thai subjects

Every subject was administered a single dose of three tablets of DHA-PQP from previous studies. To avoid unnecessary exposure of DHA-PQP again, we propose to include the results of DHA-PQP arm from these previous studies and ask the healthy subjects to participate this study for receiving only single dose of three tablet of DHA-PQP (40mg/320mg) and two tablet of Mefloquine (250mg) on first admission and single dose of two tablet of Mefloquine on second admission.

DETAILED DESCRIPTION:
Artemisinin resistance poses the greatest threat to current global initiatives to control and eliminate malaria. The World Health Organisation recommends the use of the artemisinin combination therapy (one partner drug combine with artemisinin as the back bone) (ACTs) instead of the single drug. The reduction in artemisinin sensitivity has left partner drugs within ACTs exposed too much larger number of parasites and unsurprisingly cure rates with ACTs have begun to fall substantially.

Recently, the Mahidol Oxford Tropical Medicine Research Unit (MORU) has applied for and received funding for an extension of the TRAC project. The proposed extension project, named TRACII, will further map artemisinin and partner drug resistance in the South-East Asian region. Also, TRACII aims to investigate the safety, pharmacokinetic characteristics and efficacy of a novel combination of an artemisinin-derivative and two long acting partner drugs, piperaquine and mefloquine.

It is necessary that the potential drug-drug interactions of mefloquine and dihydroartemisinin-piperaquine (DHA-PQP) are characterized. Piperaquine and Mefloquine are both metabolized by Cytochrome P450 3A4 (abbreviated CYP3A4) enzyme which potentially results in clinically significant drug-drug interactions that can cause unanticipated adverse reactions or therapeutic failures because of the suboptimal drug exposures to the parasite.

The study will evaluate the pharmacokinetic interaction and safety profile focusing on the cardiogenic effect (QTc prolongation) of this triple combinations of DHA-PQP and mefloquine. Piperaquine and Mefloquine are both metabolized by Cytochrome P450 3A4 enzyme which potentially results in clinically significant drug-drug interactions.

These safety and pharmacokinetic data will be translated to support the intervention in the Tracking Resistance to Artemisinin Collaboration II (TRACII) project.

This is an open-label sequential pharmacokinetic study in 16 healthy G6PD normal Thai subjects. The 16 subjects have participated in a healthy volunteer studies in the past either i) Open-Label Study to Evaluate Potential Pharmacokinetic Interaction of Orally Administered primaquine and dihydroartemisinin-piperaquine in Healthy Adult Subjects or ii) Comparison of the electrocardiographic effects in relation to Pharmacokinetic profile of chloroquine and piperaquine in healthy Thai subjects in which they were administered a single dose of three tablets of DHA-PQP. To avoid unnecessary exposure of other healthy subjects to this study, we propose to include the result of these previous studies and ask the healthy subjects to participate from regimen 1 and onward.

Subjects will be admitted in the inpatient ward to receive 2 drug regimens: regimen 1 (Mefloquine with DHA-PQP) and regimen 2 (Mefloquine). Every subject will have 1 screening and 2 admissions in the hospital

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as judged by a responsible physician with no abnormality identified on a medical evaluation including medical history and physical examination.
2. Males and Females non-smoker aged between 18 years to 60 years.
3. Males and Females weight between 36-75 kilograms.
4. A female is eligible to enter and participate in this study if she is:

   * of non-childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy or double oophorectomy
   * or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum follicle stimulating hormone levels >40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy
   * or of childbearing potential, has a negative serum pregnancy test at screening and prior to start the study drug in each period, and abstain from sexual intercourse or agrees to using effective contraceptive methods (e.g., intrauterine device, hormonal contraceptive drug, tubal ligation or female barrier method with spermicide) during the study until completion of the follow-up procedures
5. A male is eligible to enter and participate in this study if he: agrees to abstain from (or use a condom during) sexual intercourse with females of childbearing potential or lactating females; or is willing to use a condom/spermicide, during the study until completion of the follow-up procedures.
6. Provide a signed and dated written informed consent prior to study participation.
7. Normal electrocardiogram (ECG) with QTc <450 msec.
8. Willingness and ability to comply with the study protocol for the duration of the trial.

Exclusion Criteria:

1. Females who are pregnant, trying to get pregnant, or are lactating.
2. The subject has evidence of active substance abuse that may compromise safety, pharmacokinetics, or ability to adhere with protocol instructions.
3. A positive pre-study hepatitis B surface antigen, positive hepatitis C antibody, or positive human immunodeficiency virus-1 (HIV-1) antibody result at screening.
4. Subjects with a personal history of cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or additional risk factors for torsades de points (heart failure, hypokalemia) or with a family history of sudden cardiac death.
5. A creatinine clearance <70 mL/min as determined by Cockcroft-Gault equation:

   Creatinine clearance (CLcr (mL/min)) = (140 - age) * Wt / (72 * Scr) (multiply answer by 0.85 for females) Where age is in years, weight (wt) is in kg, and serum creatinine (Scr) is in units of mg/dL [Cockcroft, 1976].
6. History of alcohol or substance abuse or dependence within 6 months of the study.
7. Use of prescription or non-prescription drugs except paracetamol at doses of up to 2 grams/day, including vitamins, herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 times the drug half-life (whichever is longer) prior to the first dose of study medication until the completion of the follow-up procedure, unless in the opinion of investigator, the medication will not interfere with the study procedures or compromise subject safety; the investigator will take advice from the manufacturer representative as necessary.
8. The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-life, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of study medication.
9. The subject is unwilling to abstain from ingesting alcohol within 48 hours prior to the first dose of study medication until collection of the final pharmacokinetic sample during each regimen.
10. Subjects who have donated blood to the extent that participation in the study would result in more than 300 mL blood donated within a 30-day period. Note: This does not include plasma donation.
11. Subjects who have a history of allergy to the study drug or drugs of this class, or a history of drug or other allergy that, in the opinion of the investigator, contraindicates participation in the trial. In addition, if heparin is used during pharmacokinetic sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
12. Lack of suitability for participation in this study, including but not limited to, unstable medical conditions, systemic disease manifested by tendency to granulocytopenia e.g. rheumatoid arthritis and lupus erythematosus that in the opinion of the investigator would compromise their participation in the trial.
13. Aspartate transaminase (AST) or Alanine transaminase (ALT) >1.5 upper limit of normal (ULN)
14. Subjects with history of renal disease, hepatic disease, and/or cholecystectomy
15. History of antimalarial drugs use including but not limited to mefloquine, chloroquine, primaquine, artesunate, piperaquine and pyronaridine treatment within 3 months.
16. Subject who received quinacrine in last 30 days.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability parameters (including adverse events, clinical laboratory, and vital signs assessments) | approximately 4 months
  Safety and tolerability parameters, including adverse events, clinical laboratory, and vital signs assessments, in particular QTc prolongation for DHA-PQP in combination with mefloquine.
Area under the curve and maximum concentration | approximately 36 days
  Area under the concentration-time curve [AUC 0-∞ and AUC 0-last] and maximal concentration (Cmax) for mefloquine and metabolites when given alone and together with DHA-PQP.
Area under the curve and maximum concentration | approximately 36 days
  Area under the concentration-time curve [AUC0-∞ and AUC0-last] and maximal concentration (Cmax) for piperaquine and dihydroartemisinin when given alone as DHA-PQP and together with mefloquine.

SECONDARY OUTCOMES:
Pharmacokinetic parameters ((i.e. elimination clearance (CL/F), terminal elimination half-life (t1/2) and apparent volume of distribution (Vd) | approximately 36 days
  Estimate pharmacokinetic parameters (i.e. elimination clearance (CL/F), terminal elimination half-life (t1/2) and apparent volume of distribution (Vd) for mefloquine, dihydroartemisinin and piperaquine when given alone and in combination.
Genetic abnormality | approximately 4 months
  In case of any abnormal metabolisms in individuals, related genetic tests may be performed to determine if there is any genetic abnormality. Such data may be useful in predicting those who may not obtain the full therapeutic or prophylactic benefit of study drugs.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Tropical Medicine, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Hanboonkunupakarn B, van der Pluijm RW, Hoglund R, Pukrittayakamee S, Winterberg M, Mukaka M, Waithira N, Chotivanich K, Singhasivanon P, White NJ, Dondorp AM, Tarning J, Jittamala P. Sequential Open-Label Study of the Safety, Tolerability, and Pharmacokinetic Interactions between Dihydroartemisinin-Piperaquine and Mefloquine in Healthy Thai Adults. Antimicrob Agents Chemother. 2019 Jul 25;63(8):e00060-19. doi: 10.1128/AAC.00060-19. Print 2019 Aug. PMID 31182525